CLINICAL TRIAL: NCT01691235
Title: Evaluation of the SIMpill Medication Dispensing Device in the Treatment of Chronic Hepatitis C
Brief Title: SIMpill Medication Dispensing Device in the Treatment of HCV
Acronym: SIMpill HCV
Status: Withdrawn | Type: Observational
Why Stopped: No subjects enrolled due to delay in device production
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 12-1293
Record Dates: First submitted 2012-09-17; First posted 2012-09-24 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Hepatitis C Virus
Keywords: SIMpill; HCV; Chronic Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A blood draw (about 1 tablespoon) if the medication is not working for a subject. This blood draw is another way for the study team to measure adherence to the therapy. This blood draw will be taken only once at the time HCV in the blood return to high levels. This blood draw will measure HCV resistance.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm 1: Subjects in this arm will receive their medication (telaprevir, interferon and ribavirin) dispensed using the Simpill device. The study staff will have access to data from the device during therapy and will be able to give subjects feedback on adherence during the course of therapy. The study team will refill the device as the medication is needed. The device will be configured to remind a subject each time a dose is missed. Subjects in this study arm will receive a text message each time a dose of medication is missed. This message will only go to the telephone number specified by the subject and will not go to members of the study team.
  Interventions: Device: SIMpill device
- Arm 2: Subjects in this arm will receive their medication (telaprevir, interferon and ribavirin) as standard of care therapy where the SIMpill device will not be used.

INTERVENTIONS:
Device: SIMpill device — The SIMpill device is an automated pill dispensing device that records a time stamp each time the device is opened and a dose of medication is taken. This works through a computer chip that is housed inside of the pill dispensing device that is activated each time the pill box is opened. Physicians can download this data and generate a precise account of the patient's adherence to the medication dosing schedule. In addition, if a dose is missed, the SIMpill device can be set to automatically notify the patient by text message if a dose is overdue.
  Groups: Arm 1

SUMMARY:
Subjects are being asked to participate in this study because they have genotype 1 Hepatitis C Virus (HCV) and will be taking the standard of care drugs pegylated interferon, ribavirin, and telaprevir as part of their routine care. The purpose of this study is to see if the SIMpill automated pill dispensing device can help subjects take their medications at the times the doctor has instructed them to take it.

The SIMpill device is an automated pill dispensing device that records a time stamp each time the device is opened and a dose of medication is taken. Physicians can download this data and generate a precise account of when you have taken your medication. In addition, if a dose is missed, the SIMpill device can be set to automatically notify you by text message if a dose is overdue. The Simpill device is a new way to keep track of when you take your HCV medications and will also help remind you when you forget to take a dose. In addition, this information will help your doctors understand how taking medication on time effects the success of the therapy.

DETAILED DESCRIPTION:
* Patients with genotype 1 HCV who are candidates for therapy with telaprevir, pegylated interferon and ribavirin will be eligible for the study.
* All patients enrolled in this study will receive a standard of care regimen of telaprevir /pegylated interferon and ribavirin. This includes medication dosages, follow-up, and monitoring. The only exception will be the mode of medication dispensing.
* Patients will be asked to bring their Simpill devices to their regularly scheduled clinic visits at which time medication adherence information will be downloaded by study personnel. Each visit will be a regularly scheduled standard of care visit and no additional clinic visits will be needed for the patient in the Simpill study arm.
* In the event that any patient demonstrated viral breakthrough during therapy, those patients will be offered an additional blood draw to screen for viral resistance. This will be important to understand if patients using the Simpill device have better adherence to the medication regiment which results in lower incidence of viral resistance.
* Patients in the study arm will receive a text messages each time a dose of medication is missed. This message will only go to the telephone number specified by the patient and will not go to members of the study team. Patients who do not have text messaging capability will not be eligible for this study.
* The initial study will be a pilot study designed to obtain preliminary data regarding the feasibility of this device. This study is powered to detect differences in viral kinetics over the first 4 weeks.
* In the event that Vertex receives FDA approval for BID dosage of telaprevir prior to funding and initiation of the study, the most currently approved dosing (BID) will be used instead of q8 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 - 70 with genotype 1 HCV
* Compensated liver disease who are independently deemed an appropriate candidate for telaprevir containing HCV treatment regimen

Exclusion Criteria:

* Prior liver transplantation
* Co-infection with other types of viral hepatitis and HIV

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the outpatient/inpatient Liver GI clinic at the University of Chicago Medical Center
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Improved SVR Rates | 2 years
  To determine if the Simpill devise will improve viral kinetics from week 0 to week 4, leading to improved SVR rates.

SECONDARY OUTCOMES:
Improved Patient Adherence Rates | 2 years
  To determine overall adherence rates among patients taking telaprevir

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Aronsohn, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States